CLINICAL TRIAL: NCT01426906
Title: A Randomized, Open-Label, Drug-Drug Interaction Study To Evaluate The Effect Of Ketoconazole Or Rifampicin On The Pharmacokinetic Characteristics And Safety Of Lc15-0444 In Healthy Male Volunteers
Brief Title: Pharmacokinetic Drug Interaction Study in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LG-DPCL007
Record Dates: First submitted 2011-08-31; First posted 2011-09-01 (Estimated); Last update posted 2011-09-01 (Estimated); Status verified 2011-08

CONDITIONS: Healthy Male Volunteers
MeSH Terms: interventions — Ketoconazole; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study A (Experimental)
  Interventions: Drug: Ketoconazole
- Study B (Experimental)
  Interventions: Drug: rifampicin

INTERVENTIONS:
Drug: Ketoconazole — Period 1 : LC15-0444 Period 2 : LC15-0444 with ketoconazole
  Arms: Study A
Drug: rifampicin — Period 1 : LC15-0444 Period 2 : LC15-0444 with rifampicin
  Arms: Study B

SUMMARY:
A Randomized, Open Label, Drug-Drug interaction study to investigate effect of ketoconazole or rifampicin on the Pharmacokinetic characteristics and safety of LC15-0444 in Healthy Male Volunteers.

DETAILED DESCRIPTION:
This study is a randomized, open-label, 2-period, 3-treatment, 1-sequence, drug-drug interaction study in healthy volunteers to evaluate effect of ketoconazole or rifampicin on the PK characteristic and safety of LC15-0444.

Eligibility for participation of this study will be determined by demographic information, medical history, physical examination, electrocardiogram (ECG) and clinical laboratory tests within 4 weeks(-28 d ~ -2 d) before the first drug administration(1 d). Eligible subjects will be randomized to one of study treatment groups.

According to the characteristics of anti-diabetic drugs, it is expected to be administered with other drugs in many patients. Therefore, Drug-Drug Interaction with CYP3A4 inducer and inhibitor should be identified in this trial.

ELIGIBILITY:
Inclusion Criteria:

* Is a healthy male between 20 and 50 years old
* Has BMI result between 19 and 26 kg/m2 at screening; and a total body weight over 55 kg. BMI(kg/m2) = body weight(kg)/{height(m)}2.
* Is willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures
* Agrees to use an adequate means of contraception during clinical trials

Exclusion Criteria:

* Subjects with evidence or history of clinically significant hepatic, renal, digestive, neurologic, pulmonary, musculoskeletal, endocrine, hematological, cardiovascular or psychiatric disease
* Subjects with evidence or history of gastrointestinal disease or surgery possibly affecting drug absorption.
* Subjects with history of hypersensitivities or clinically significant adverse events caused by DPPIV inhibitors, ketoconazole, rifampicin, and other drugs
* Subjects who have donated a unit of blood within 60 days or blood components within 30 days before the first administration of the investigational product.
* Subjects who consume excessive alcohol or caffeine; who excessively smoke

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Cmax | Until Day 18 or 20
AUC(last) | Until Day 18 or 20
AUC(0-24hr) | Until Day 18 or 20
Tmax | Until Day 18 or 20
t(1/2beta) | Until Day 18 or 20
(6-b-hydrocortisol)/(cortisol) ratio | Until Day 20

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Noh YH, Lim HS, Jin SJ, Kim MJ, Kim YH, Sung HR, Choi HY, Bae KS. Effects of ketoconazole and rifampicin on the pharmacokinetics of gemigliptin, a dipeptidyl peptidase-IV inhibitor: a crossover drug-drug interaction study in healthy male Korean volunteers. Clin Ther. 2012 May;34(5):1182-94. doi: 10.1016/j.clinthera.2012.04.001. Epub 2012 Apr 24. PMID 22534255